CLINICAL TRIAL: NCT02263859
Title: ImThera Medical Targeted Hypoglossal Neurostimulation Study #3
Brief Title: Targeted Hypoglossal Neurostimulation Study #3
Acronym: THN3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ImThera Medical, Inc. (Industry)
Collaborators: LivaNova (Industry)
Responsible Party: Sponsor
Organization: LivaNova (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMT 2014-01
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): The Treatment Group will be implanted with the aura6000 System and have therapy turned ON at the Month 1 follow-up visit.
  Interventions: Device: aura6000 System
- Control (Other): The Control Group will be implanted with the aura6000 System and receive treatment as-usual, (i.e. any non-PAP, non-surgical OSA treatment including oral appliances and positional devices being used prior to enrollment in the study) until 14 days (washout period) prior to the Month 4 visit. At the Month 4 + 1 day follow-up visit, subjects in the Control Group will have therapy turned ON for the duration of the study.
  Interventions: Device: aura6000 System

INTERVENTIONS:
Device: aura6000 System — The aura6000 System is intended to unilaterally stimulate the hypoglossal nerve which innervates the muscles of the tongue. The aura6000 System stimulates the hypoglossal nerve cyclically and continuously during sleep to maintain muscle tone of the tongue and upper airway during sleep. Stimulation is generated by a programmable, multi-current source, implantable neurostimulator (IPG) and delivered to the hypoglossal nerve by a lead with multi-contact cuff electrode (lead).
  Other Names: THN Therapy; ImThera Medical

SUMMARY:
The purpose of this study is to evaluate the benefits and risks of hypoglossal nerve stimulation with the ImThera Medical aura6000 System as a potential therapeutic option for individuals with moderate to severe OSA that have failed or do not tolerate PAP.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the safety and effectiveness of the aura6000 System for the treatment of moderate to severe obstructive sleep apnea (OSA) in individuals who have failed or do not tolerate positive airway pressure (PAP) therapy or have failed or are intolerant of or refuse indicated alternative OSA treatments (such as oral appliances, positional devices and conventional sleep surgeries). PAP failure is defined as an inability to eliminate OSA (AHI > 20 despite PAP usage) and PAP intolerance is defined as: 1) inability to use PAP (greater than 5 nights per week of usage; usage defined as greater than 4 hours of use per night); or 2) unwillingness to use PAP (for example, a patient returns the PAP system after attempting to use it). The results of this study are anticipated to provide reasonable assurance of the safety and effectiveness of the aura6000 System when used as intended and to support the application for FDA Premarket Approval of the system.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Individual has failed or does not tolerate PAP therapy
* Has failed or refuses alternative OSA treatments (e.g.surgery, oral appliances, and behavioral treatments)
* AHI ≥ 20 (Moderate to severe OSA)

Exclusion Critera:

* Implanted with another active implantable device
* Body mass index (BMI) ≥ 35 kg/m²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Improvement in Apnea Hypopnea Index (AHI) | Baseline to 4 months post-implant
  Proportion of subjects who experience improvement in the apnea-hypopnea index (AHI) at the Month 4 visit as defined above in the AHI Responder definition.
  It is hypothesized that the observed responder rate in the Treatment Group will be significantly greater than the responder rate in the Control Group at 4 months post-implant.
Improvement in Oxygen Desaturation Index (ODI) | Baseline to 4 months post-implant
  Proportion of subjects who experience improvement in the oxygen desaturation index 4% (ODI 4%) at the Month 4 visit as defined above in the ODI Responder definition.
  It is hypothesized that the observed responder rate in the Treatment Group will be significantly greater than the responder rate in the Control Group at 4 months post-implant.
Safety Analysis | Baseline to 12 months post-implant
  Estimate the incidence of serious adverse events (SAEs) related to the aura6000 device or procedure, including any unanticipated adverse device effects.

SECONDARY OUTCOMES:
Long-term Responder Rate | Baseline to 12 months post-implant
Change in Epworth Sleepiness Scale (ESS) | Baseline to 4 months post-implant
Change in Functional Outcomes of Sleep (FOSQ) | Baseline to 4 months post-implant
Change in EuroQol 5 Dimensional (EQ-5D) | Baseline to 4 months post-implant

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Schwartz, MD, Principal Investigator — Professor (ret.), Johns Hopkins University
Locations (20):
- United States (14):
  - ENT Associates of San Diego, Chula Vista, California
  - Tower ENT, Los Angeles, California
  - SENTA Clinic, San Diego, California
  - Ear, Nose, and Throat Associates of South Florida, Boca Raton, Florida
  - Morton Plant Mease Healthcare, Safety Harbor, Florida
  - Advanced ENT Asociates, Atlanta, Georgia
  - Center for ENT and Allergy, Carmel, Indiana
  - Kentucky Research Group, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - ENT and Allergy Associates, New York, New York
  - Intrepid Research, Cincinnati, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Methodist Physicians, Memphis, Tennessee
  - FutureSearch Trials, Austin, Texas
- Clinique Univ. Saint-Luc, Brussels, Belgium
- France (2):
  - Pitie Salpetriere, Paris
  - Foch Hospital, Suresnes
- Ruprechts-Karls University, Mannheim, Germany
- Bnai Zion Medical Center, Haifa, Israel
- Hospital CUF Porto, Porto, Portugal

REFERENCES:
- [Derived] Schwartz AR, Jacobowitz O, Eisele DW, Mickelson SA, Miller MB, Oliven A, Certal V, Hopp ML, Winslow DH, Huntley TC, Nachlas NE, Pham LV, Gillespie MB, Weeks BH, Lovett EG, Shen J, Malhotra A, Maurer JT. Targeted Hypoglossal Nerve Stimulation for Patients With Obstructive Sleep Apnea: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2023 Jun 1;149(6):512-520. doi: 10.1001/jamaoto.2023.0161. PMID 37022679